CLINICAL TRIAL: NCT02157883
Title: A Phase I, Open-label, Non-randomised Study to Assess the Effect of Itraconazole (a CYP3A4 Inhibitor) on the Pharmacokinetics of a Single Oral Dose of AZD9291 in Patients With EGFRm Positive NSCLC Whose Disease Has Progressed on an EGFR TKI
Brief Title: Study to Assess the Effect of Itraconazole (a CYP3A4 Inhibitor) on the Pharmacokinetics of AZD9291, in Patients With EGFR Positive Non-small Cell Lung Cancer. Patients Will be Chosen From Those Who Have Already Been Prescribed an EGFR TKI Medicine (Such as Iressa or Tarceva)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Other
Other Study IDs: D5160C00012; 2014-001557-16 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Non Small Cell Lung Cancer; Advanced (Inoperable) Non Small Cell Lung Cancer
Keywords: oncology, cancer, non small cell lung cancer, anticancer drug, pharmacokinetics, AZD9291, intraconazole, EGFR sensitivity mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — osimertinib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 alone, AZD9291+itraconozole (Experimental): Sequential treatments of AZD9291 alone followed by AZD9291+itraconazole, with a washout period in between.
  Interventions: Procedure: Pharmacokinetic sampling; Drug: AZD9291; Drug: Itraconazole

INTERVENTIONS:
Procedure: Pharmacokinetic sampling — Blood samples taken pre and post dosing with AZD9291+/- itraconazole
Drug: AZD9291 — AZD9291 tablets: Part A 80mg od, days 1 and 10 only. Part B 80mg od for 12 months.
Drug: Itraconazole — Itraconazole tablets: 2x100mg bd, Part A days 6 to 19 only

SUMMARY:
This is a 2 part study in patients with EGFRm+ non small cell lung cancer (NSCLC), whose disease has progressed on an EGFRm TKI, who are refractory or resistant to standard therapy. Part A will assess the effect of multiple oral doses of itraconazole on the single dose pharmacokinetic (PK) parameters of AZD9291. On completion of Part A, patients may continue to take AZD9291 tablets (Part B) following the collection of the 216 hour sample on Day 19 if they and the Investigator deem it appropriate, until such time as their disease progresses, the Investigator believes they are no longer deriving clinical benefit, or they stop taking AZD9291 for any other reason

ELIGIBILITY:
For inclusion in the study, patients should fulfil the following criteria:

1. Male or female, aged at least 18 years.
2. Histological or cytological confirmation diagnosis of NSCLC.
3. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, eg, gefitinib or erlotinib. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
4. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
5. ECOG performance status 0-1 with no deterioration over the previous 2 weeks.
6. Patients must have a life expectancy of ≥12 weeks as estimated at the time of screening.
7. Evidence of non-childbearing status for women of childbearing potential, or post-menopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of Part A, or post menopausal status. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; women under 50 years old would be consider postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution; documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
8. Male patients should be willing to use barrier contraception, ie, condoms, until 6 months after last study drug is taken.

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
2. Treatment with any of the following: Treatment with an EGFR TKI w/in 8 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment; Any cytotoxic chemotherapy, investigational agents or other anticancer drugs w/in 14 days of the first dose of study treatment; Major surgery (excluding placement of vascular access) within 4 weeks of the first dose; Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment; Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP2C8 and of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4, CYP2C8, and/ or CYP1A2.
3. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the end of Part A.
5. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: ANC <1.5 x 10^9/L; Platelet count <100 x 10^9/L; Haemoglobin <90 g/L; ALT >2.5 x the institutional ULN if no demonstrable liver metastases or >5 x institutional ULN in the presence of liver metastases; AST >2.5 x institutional ULN if no demonstrable liver metastases or >5 x institutional ULN in the presence of liver metastases; Total bilirubin >1.5 x institutional ULN if no liver metastases or >3 x institutional ULN in the presence of documented Gilbert's Syndrome or liver metastases; Creatinine >1.5 x institutional ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft-Gault formula); confirmation of creatinine clearance is only required when creatinine is >1.5 x institutional ULN.
8. Any of the following cardiac criteria: Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) >450 msec obtained from 3 ECGs; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec; Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
9. Patients unable to swallow oral medication or patients with GI disorders or significant GI resection likely to interfere with the absorption of AZD9291.
10. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
11. Women who are breastfeeding.
12. Patients with a known hypersensitivity to AZD9291 or itranconazole or any of their excipients.

12. Concomitant medication contraindicated for use with itraconazole (including, but not limited to): cisapride, oral midazolam, nisoldipine, pimozide, quinidine, dofetilide, triazolam, levacetylmethadol (levomethadyl), 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG-CoA)- reductase inhibitors metabolized by CYP3A4, such as lovastatin and simvastatin, ergot alkaloids metabolized by CYP3A4, such as dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine).

13. For optional genetic research: Previous allogenic bone marrow transplant or non-leukocyte depleted whole blood transfusion within 120 days of sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (13):
- United States (2):
  - Research Site, San Diego, California
  - Research Site, Cleveland, Ohio
- Belgium (2):
  - Research Site, Edegem
  - Research Site, Ghent
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Rotterdam
- South Korea (3):
  - Research Site, lJongno-gu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Research Site, Taipei, Taiwan
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Vishwanathan K, Dickinson PA, So K, Thomas K, Chen YM, De Castro Carpeno J, Dingemans AC, Kim HR, Kim JH, Krebs MG, Chih-Hsin Yang J, Bui K, Weilert D, Harvey RD. The effect of itraconazole and rifampicin on the pharmacokinetics of osimertinib. Br J Clin Pharmacol. 2018 Jun;84(6):1156-1169. doi: 10.1111/bcp.13534. Epub 2018 Mar 23. PMID 29381826
- See also: StudyD5160C00012 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2989&filename=StudyD5160C00012_redacted.pdf
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00012&attachmentIdentifier=7962822a-61ed-4153-820b-32dcdea4f6c2&fileName=D5160C00012_study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 6 November 2014; Last Subject Last Visit Part A: 3 April 2015 and Part B: 31 March 2016. Study performed at 15 sites across Asia, North America and Western Europe. Part A assessed effect of multiple doses of itraconazole on PK of AZD9291; Part B allowed subjects further access to AZD9291 and provided additional safety data.
Pre-assignment Details: The 39 patients started Period 1 and received treatment.
Groups:
- AZD9291 and Itraconozole (Part A); AZD9291 Alone (Part B): In Part A of the study, sequential treatments of AZD9291 alone (including a washout) followed by AZD9291+itraconazole. Each patient received single 80 mg oral doses of AZD9291 tablets on Days 1 and 10, and in addition received itraconazole capsules 200 mg twice daily on Days 6 to 18.
  In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Period: Part A: Day 1-5 (AZD9291 Alone)
Arm/Group | AZD9291 and Itraconozole (Part A); AZD9291 Alone (Part B)
Started | 39
Completed | 38
Not Completed | 1
Period: Part A: Day 6-18 (AZD9291+Itraconozole)
Arm/Group | AZD9291 and Itraconozole (Part A); AZD9291 Alone (Part B)
Started | 39
Completed | 38
Not Completed | 1
Not completed — Adverse Event | 1
Period: Part B: Day 19 to End Part B (AZD9291)
Arm/Group | AZD9291 and Itraconozole (Part A); AZD9291 Alone (Part B)
Started | 38
Completed | 16
Not Completed | 22
Not completed — Adverse Event | 3
Not completed — Disease progression | 15
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | AZD9291 and Itraconozole (Part A); AZD9291 Alone (Part B)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of maximum plasma AZD9291 concentration
Time Frame: Blood samples collected on Day 1 and Day 10 at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, and 216 hours post AZD9291 dose in Part A.
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine outcome measure without important protocol deviations/violations and excluding Period 2 data for patients meeting carry-over exclusion criterion (defined as Period 2 pre-dose concentration >10% of Cmax).
Measure: Geometric Mean (Full Range); unit: nM
Groups:
- AZD9291 Alone: Single oral dose of 80mg AZD9291 on Day 1
- AZD9291+Itraconazole: Single oral dose 80mg AZD9291 on Day 10, itraconazole 200mg twice daily dosing on Days 6-18
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 30
nM | 242.5 [88.8 to 704] | 201.7 [78.2 to 676]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; Study sized so experiment-wise power for the upper bound of the 90% CIs of geometric mean ratios for both AUC and Cmax of AZD9291 being below 200% was 90% (95% for each parameter). Within patient CV assumed to be 34%. A 50% increase in exposure was also assumed; Test type: Non-Inferiority or Equivalence — Upper bound of the 90% CIs below 200%; Geometric mean ratio = 79.87, 90% CI 2-sided [73.15 to 87.21] — AZD9291+itraconazole / AZD9291 alone. Results based on linear mixed-effects model with treatment as fixed effect and patient as a random effect

2. Primary Outcome: AUC of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 33 | 30
nM*h | 13520 [6510 to 40400] | 17090 [7130 to 59600]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Upper bound of the 90% CIs below 200%; Geometric mean ratio = 124.17, 90% CI 2-sided [114.61 to 134.53] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC(0-120) of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration time curve from zero to 120 hours
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 31
nM*h | 10280 [4980 to 27500] | 11370 [5100 to 37500]

4. Secondary Outcome: AUC(0-t) of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of area under the plasma concentration curve from time zero to last quantifiable dose
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 31
nM*h | 12260 [6090 to 33600] | 14520 [6280 to 49600]

5. Secondary Outcome: Tmax of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of time to Cmax
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 30
hours | 4.00 [2.03 to 11.87] | 6.04 [3.00 to 72.00]

6. Secondary Outcome: t1/2 of AZD9291
Description: Pharmacokinetics of AZD9291 by assessment of the terminal half-life
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 30
hours | 61.05 [38.7 to 131] | 78.36 [56.3 to 150]

7. Secondary Outcome: CL/F of AZD9291
Description: Rate and extent of absorption of AZD9291 by assessment of apparent clearance following oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 33 | 30
L/h | 11.84 [3.96 to 24.6] | 9.368 [2.69 to 22.5]

8. Secondary Outcome: Vz/F of AZD9291
Description: Rate and extent of absorption of AZD9291 by assessment of the apprarent volume of distribution
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 33 | 30
L | 1019 [491 to 2310] | 1059 [344 to 2630]

9. Secondary Outcome: Cmax of AZ5104
Description: Pharmacokinetics of AZ5104 (metabolite to AZD9291) by assessment of maximum plasma AZ5104 concentration
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine outcome measure without important protocol deviations/violations and excluding Period 2 data for patients meeting carry-over exclusion criterion (defined as Period 2 pre-dose AZ5104 concentration >20% of Cmax).
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 16
nM | 8.568 [2.36 to 23.4] | 5.746 [2.15 to 15.8]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 75.87, 90% CI 2-sided [64.18 to 89.69] — AZD9291+itraconazole / AZD9291 alone. No pre-specified margins for equivalence test for metabolites, but analysed for consistency with AZD9291 analysis

10. Secondary Outcome: AUC of AZ5104
Description: Pharmacokinetics of AZ5104 (metabolite to AZD9291) by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 31 | 15
nM*h | 1155 [367 to 4360] | 941.4 [337 to 2620]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 108.25, 90% CI 2-sided [94.36 to 124.19] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Cmax of AZ7550
Description: Pharmacokinetics of AZ7550 (metabolite to AZD9291) by assessment of maximum plasma AZ7550 concentration
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine outcome measure without important protocol deviations/violations and including Period 2 data (since all patients met carry over criteria of Period 2 pre-dose AZ7550 concentration >20% of Cmax).
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 34 | 33
nM | 4.321 [1.64 to 11.7] | 1.897 [0.659 to 5.42]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 44.33, 90% CI 2-sided [39.94 to 49.21] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: AUC of AZ7550
Description: Pharmacokinetics of AZ7550 (metabolite to AZD9291) by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of AZD9291 and had sufficient postdose PK assessments to determine outcome measure without important protocol deviations, where AUC possible to calculate, and including Period 2 data (all patients met carry over criteria of Period 2 pre-dose AZ7550 concentration >20% of Cmax).
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 Alone | AZD9291+Itraconazole
Number analyzed (Participants) | 33 | 19
nM*h | 624.1 [210 to 1700] | 292.1 [158 to 578]
Statistical Analysis 1: Comparison: AZD9291 Alone vs AZD9291+Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 49.02, 90% CI 2-sided [43.70 to 54.99] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 3 weeks for Part A; up to approximately 15.5 months for Part B and approximately 16 months for Overall (Parts A and B combined).
Description: Part A: Adverse events (AEs) collected from day of first dose until day prior to first dose in Part B (Day 19), or until 30 days after last dose if discontinued in Part A. Part B: AEs collected from day of first dose in Part B until 30 days after last dose, or until last dose in Part B for those entering continued access phase (CAP).
Groups:
- Overall: Parts A and B of the study combined.
- Part A: In Part A of the study, each patient received a single 80 mg oral AZD9291 tablet dose in each of 2 treatment periods (AZD9291 dosing on Days 1 and 10). Patients additionally received itraconazole 200 mg twice daily dosing from Days 6 to 18.
- Part B: In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Arm/Group | Overall | Part A | Part B
Serious Adverse Events (participants affected / at risk) | 12/39 | 3/39 | 9/38
Other Adverse Events (participants affected / at risk) | 39/39 | 24/39 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=39) | Part A (N=39) | Part B (N=38)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Hepatic enzyme increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=39) | Part A (N=39) | Part B (N=38)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9) | 2 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 2 (2) | 13 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (18) | 7 (8) | 10 (10)
Oesophageal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 10 (15) | 6 (8) | 6 (7)
Fatigue (General disorders) | 12 (13) | 3 (3) | 9 (10)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 4 (5) | 2 (2) | 3 (3)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 8 (9) | 0 (0) | 8 (9)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (5) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (8) | 0 (0) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 0 (0) | 4 (9)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 0 (0) | 3 (4)
Blood creatine increased (Investigations) | 2 (3) | 0 (0) | 2 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (4) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 1 (1) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 7 (9) | 4 (4) | 3 (5)
Headache (Nervous system disorders) | 7 (9) | 1 (1) | 6 (8)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1) | 3 (3)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
At end of Part B, the CAP allowed patients to continue receiving AZD9291 if still deriving clinical benefit. No clinical data was databased during the CAP; thus AE data is presented to end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.